CLINICAL TRIAL: NCT03351725
Title: Incidence of Peripheral Intravenous Cannula Colonization in a Swedish County Hospital
Brief Title: Peripheral Venous Catheter Colonization Study
Acronym: IPICCS
Status: Completed | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Boel Andersson Gäre, Professor, Linkoeping University
Other Study IDs: 0709323371
Record Dates: First submitted 2017-11-15; First posted 2017-11-24 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Catheters, Indwelling; Catheter-Related Infections
Keywords: peripheral venous catheter; catheter colonization
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripheral venous catheter indwell time more than 48 hours
  Interventions: Device: peripheral venous catheter (PVC)

INTERVENTIONS:
Device: peripheral venous catheter (PVC) — No intervention is made only in situ swab from the PVC

SUMMARY:
Peripheral intravenous cannulas (PIVCs) are utilized in large scale in modern health care. Known complications due to a PIVC are phlebitis, thrombosis, bleeding, nerve damage and infection. PIVC-related infection causes morbidity, mortality and increased healthcare costs. PIVC-related infections can and should be prevented.

Indwell time is a known risk factor for PIVC-related infection. Another factor potentially influencing the risk of developing PIVC-related infection is what type of PIVC that is being used. Roughly there are two types of PIVCs. One with an open injection valve and another with a closed injection valve. The former being far more used in our hospital and the latter being suggested as lowering the risk of PIVC-related infection compared to the open one.

The investigators aim with this study is to evaluate the incidence of PIVC-colonization in 300 patients at our 500-bed secondary level hospital in Sweden, as a first step in trying to understand what healthcare-providers can improve regarding prevention of PIVC-related infections.

DETAILED DESCRIPTION:
Background:

Peripheral intravenous cannulas (PIVCs) are utilized in large scale in modern health care. Known complications due to a PIVC are phlebitis, thrombosis, bleeding, nerve damage and infection. PIVC-related infection causes morbidity, mortality and increased healthcare costs. In an Australian study the investigators found the presence of a PIVC the most frequent cause (36%) of healthcare-associated Staphylococcus aureus bacteraemia during 2012. PIVC-related infections can and should be prevented.

Indwell time is a known risk factor for PIVC-related infection. Another factor potentially influencing the risk of developing PIVC-related infection is what type of PIVC that is being used. Roughly there are two types of PIVCs. One with an open injection valve and another with a closed injection valve. The former being far more used in Ryhov County Hospital, Sweden, and the latter being suggested as lowering the risk of PIVC-related infection compared to the open one.

In a systematic review from 2006 Maki et al report a point incidence of blood stream infections of 0,5 per 1000 catheter-days in PIVCs. In 2014 Hammarskjöld reported an incidence of 0,6 per 1000 catheter-days regarding central venous catheters (CVC). Maki et al concludes "…, infection control programs must strive to consistently apply essential control measures and preventive technologies with all types of intravascular devices." The investigators find there is a gap between the large scale utilization of PIVCs and the knowledge about PIVC-related infections and recommendations on how to prevent them. Hammarskjöld et al has done research on infections related to CVCs, subcutaneous venous ports and on arterial cannulas but not PIVCs.

The aim with this study is to evaluate the incidence of PIVC-colonization at Ryhov County Hospital, a 500-bed secondary level hospital in Sweden, as a first step in trying to understand what can be done to improve work regarding prevention of PIVC-related infections.

Materials and methods

Setting The hospital is a 500-bed general county hospital including most medical, oncological and surgical specialties except neurosurgery and cardiac surgery. No solid organ or stem cell transplantations are performed.

Patients Patients admitted to surgical, medical or infectious wards were regularly included by a specifically trained nurse from June 2016 until December 2017.

Inclusion criteria: Patients ≥ 18 years of age with a PIVC in situ for 48 hours or more informed verbally and in written and invited to take part in the study. Exclusion criteria: Patients < 18 years of age.

Microbiological methods Intraluminal hub culturing from the two injection sites of the PIVC performed with sterile cotton-tipped applicators moistened with sterile sodium chloride 0,9 %. Swabs transported in Amies medium with charcoal. Identification performed by standard methods at our local microbiology laboratory (www.srga.org.accessed _ http:// www.srga.org.accessed/ _ January 1, 2007).

Statistics Descriptive. How many positive cultures and which type of microbes were found.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older hospitalized in Ryhov County Hosptial, Sweden, with perhiperal venous catheter in situ for 48 hours or more.

Exclusion Criteria:

* Under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Setting The hospital is a 500-bed general county hospital including most medical, oncological and surgical specialties except neurosurgery and cardiac surgery. No solid organ or stem cell transplantations are performed. Patients Patients admitted to surgical, medical or infectious wards were regularly included by a specifically trained nurse from June 2016 until December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Positive culture | 2-7 days
  Swab from peripheral venous catheter (PVC) in situ on patient having had the PVC for 48 hours or more.

CONTACTS AND LOCATIONS:
Overall Officials: Boel Andersson Gäre, Professor, Principal Investigator — Linkoeping University, Sweden
Locations (1):
- Ryhov County Hospital, Jönköping, Småland, Sweden

IPD SHARING:
Plan to Share IPD: No
No individual data, but the the data regarding positive Cultures and what type of microbia found will be official

REFERENCES:
- [Result] Rhodes D, Cheng AC, McLellan S, Guerra P, Karanfilovska D, Aitchison S, Watson K, Bass P, Worth LJ. Reducing Staphylococcus aureus bloodstream infections associated with peripheral intravenous cannulae: successful implementation of a care bundle at a large Australian health service. J Hosp Infect. 2016 Sep;94(1):86-91. doi: 10.1016/j.jhin.2016.05.020. Epub 2016 Jun 7. PMID 27346623
- [Result] Gonzalez Lopez JL, Arribi Vilela A, Fernandez del Palacio E, Olivares Corral J, Benedicto Marti C, Herrera Portal P. Indwell times, complications and costs of open vs closed safety peripheral intravenous catheters: a randomized study. J Hosp Infect. 2014 Feb;86(2):117-26. doi: 10.1016/j.jhin.2013.10.008. Epub 2013 Dec 1. PMID 24373830
- [Result] Maki DG, Kluger DM, Crnich CJ. The risk of bloodstream infection in adults with different intravascular devices: a systematic review of 200 published prospective studies. Mayo Clin Proc. 2006 Sep;81(9):1159-71. doi: 10.4065/81.9.1159. PMID 16970212
- [Result] Hammarskjold F, Berg S, Hanberger H, Taxbro K, Malmvall BE. Sustained low incidence of central venous catheter-related infections over six years in a Swedish hospital with an active central venous catheter team. Am J Infect Control. 2014 Feb;42(2):122-8. doi: 10.1016/j.ajic.2013.09.023. PMID 24485369
- [Result] Mermel LA. Short-term Peripheral Venous Catheter-Related Bloodstream Infections: A Systematic Review. Clin Infect Dis. 2017 Oct 30;65(10):1757-1762. doi: 10.1093/cid/cix562. PMID 29020252
- [Derived] Juhlin D, Hammarskjold F, Mernelius S, Taxbro K, Berg S. Microbiological colonization of peripheral venous catheters: a prospective observational study in a Swedish county hospital. Infect Prev Pract. 2021 Jun 7;3(3):100152. doi: 10.1016/j.infpip.2021.100152. eCollection 2021 Sep. PMID 34458717